CLINICAL TRIAL: NCT02080377
Title: A Feasibility Study Looking at the Use of Glibenclamide and metfoRmin Versus stAndard Care in gEstational diabeteS
Acronym: GRACES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRACES; 2013-004706-25 (EudraCT Number)
Record Dates: First submitted 2014-02-11; First posted 2014-03-06 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy; Gestational Diabetes
Keywords: Pregnancy; Gestational diabetes; Glycaemic control; Metformin
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glyburide; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current Standard Care (Active Comparator): Insulin + Metformin
  Interventions: Drug: Insulin
- Treatment (Active Comparator): Glibenclamide + Metformin
  Interventions: Drug: Glibenclamide

INTERVENTIONS:
Drug: Glibenclamide
  Arms: Treatment
Drug: Insulin
  Arms: Current Standard Care

SUMMARY:
The aim of this open label feasibility study is to determine recruitment rates to a randomised trial of glibenclamide compared with insulin (both in addition to maximum tolerated metformin) for the treatment of Gestational Diabetes Mellitus (GDM). This feasibility trial will inform the design of a future substantive multicentre trial to test the hypothesis that combination therapy with glibenclamide and metformin could reduce the number of pregnant women with GDM who require insulin and would be superior to metformin and insulin in terms of acceptability and cost effectiveness.

Women with GDM who have "failed" monotherapy with metformin will be recruited and randomised to either receive glibenclamide (test arm) or standard care with insulin, both in addition to their maximum tolerated dose of metformin. Patients will be recruited from three of the antenatal clinics.

This is a feasibility study in preparation for a large multicentre randomised trial to test the hypothesis that the addition of glibenclamide to metformin (combination therapy) could reduce the number of pregnant women with gestational diabetes mellitus requiring insulin, without compromising glycaemic control or other clinical outcomes. The investigators hypothesise that combination therapy with metformin and glibenclamide is likely to be preferable to metformin and insulin in terms of acceptability and cost.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with gestational diabetes who fail to achieve "adequate glycaemic control" on maximum tolerated dose metformin
* Inadequate glycaemic control is defined according to the SIGN 116 guidelines.

Exclusion Criteria:

* Pregnant women requiring insulin prior to 20 weeks gestation or after 36 weeks gestation.
* Pregnant women not taking at least 500mg metformin daily.
* Patients with suspected Type 1 diabetes mellitus presenting in pregnancy.
* Women with allergies to either glibenclamide or insulin or any of their excipients.
* Women with any contraindications to sulfonylurea therapy.
* Women unable to give informed consent.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of women willing to be randomised | 2 years
  * Retention - proportion of women randomised who remain in the study to provide outcomes
  * Adherence - proportion of clinicians who adhere to the treatment regimen(s)

SECONDARY OUTCOMES:
Glycaemic control | 2 weekly
  Safety - number of hypoglycaemic episodes needing treatment, any other adverse events
Patient satisfaction | 36-38 weeks gestation
  assessed by visual analogue scale
Clinical outcomes | 36 weeks
  Change in maternal weight between booking and 36 weeks
Clinical outcome | 40 weeks
  Mode and gestation of delivery.
Clinical Outcome | 40 weeks
  Birthweight centile (adjusted for sex and gestation at birth)
Clinical Outcome | 2 days
  Incidence of neonatal hypoglycaemia (defined as any of the following: blood glucose <2.6 mmol/l) in first 48hrs age, or given intravenous glucose or any other drug to increase blood glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Norman, MD, Principal Investigator — University of Edinburgh
Locations (5):
- United Kingdom (5):
  - Queen Elizabeth Hospital, Glasgow, Glasgow
  - Princess Royal Infirmary, Glasgow, Lanarkshire
  - Simpson Centre for Reproductive Health, Royal Infirmary Hospital, Edinburgh, Edinburgh, Lothian
  - Western General Hospital, Edinburgh, Lothian
  - St Johns Hospital, Livingston, West Lothian

REFERENCES:
- [Derived] Reynolds RM, Denison FC, Juszczak E, Bell JL, Penneycard J, Strachan MWJ, Lindsay RS, Alexander CI, Love CDB, Whyte S, Mackenzie F, Stenson B, Norman JE. Glibenclamide and metfoRmin versus stAndard care in gEstational diabeteS (GRACES): a feasibility open label randomised trial. BMC Pregnancy Childbirth. 2017 Sep 22;17(1):316. doi: 10.1186/s12884-017-1505-3. PMID 28938877